CLINICAL TRIAL: NCT03250143
Title: A Randomised Study to Assess and Compare the Efficacy of Cyclosporine Versus Azathioprine in the Treatment of Chronic Refractory Urticaria
Brief Title: To Assess and Compare the Efficacy of Cyclosporine Versus Azathioprine in the Treatment of Chronic Refractory Urticaria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Davinder Parsad, DParsad(professor), Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2017/609
Record Dates: First submitted 2017-05-19; First posted 2017-08-15 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Chronic Refractory Urticaria
MeSH Terms: interventions — levocetirizine

STUDY DESIGN:
Intervention Model Description: Randomized prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Oral cyclosporine 3mg/kg/day (200mg/day) will be started.If there is no improvement in 1 week then escalating the dose maximum upto 5mg/kg/day.
  Interventions: Drug: cyclosporine vs azathioprine
- group B (Active Comparator): Oral azathioprine will be started at 1mg/kg/day.If there is no improvement in 1 week then escalating the dose maximum upto 100mg/day
  Interventions: Drug: cyclosporine vs azathioprine

INTERVENTIONS:
Drug: cyclosporine vs azathioprine — Group A cyclosporine 3mg/kg/day and group B azathioprine 1mg/kg/day
  Other Names: levocetrizine

SUMMARY:
Fifty six patients of CRU attending the urticaria clinic in the department of Dermatology, Venereology and Leprology at the Post Graduate Institute of Medical Education and Research, Chandigarh will be recruited in the study calculated by using equivalence analysis assuming power of 90%, significance level of 5% and standard deviation of 1 and adjusting 5% of expected drop-outs after taking written informed consent. This study is undertaken with an intention to treat the patients of chronic refractory urticaria completely. Patients will be randomized into two groups A and B using computer generated random number tables, group A will receive Cyclosporine and group B will receive Azathioprine; wherein, 28 random single and double-digit numbers from 1-56 will be selected before recruitment, and patients coming on these numbers will be randomized in a particular group. Random number generation, recruitment and randomization, were all done by the same investigator..

DETAILED DESCRIPTION:
Available definition for chronic refractory urticaria (CRU) is chronic spontaneous urticaria, with disease duration of at least 6 months or above, which is not controlled with four fold increased dosage of antihistamines (as per EAACI guidelines), given for at least three consecutive months and requiring repeated courses of oral corticosteroids. There is no strict number of oral corticosteroids intake courses before the patient can be labeled as chronic refractory urticaria.

Study end- points

1. Primary end-point :

   Change in urticaria activity score (UAS7) i.e decrease more than 75% from baseline to week 12 (at end of treatment) within group A and B and comparison between corresponding groups.
2. Secondary end-points :

   1. Change in outcome scoring scale (OSS) from baseline to week 12 within group A and B.
   2. Change in UAS7 and OSS from baseline to week 24 (end of follow-up) within group A and B.
   3. Change in ASST, APST, IgE levels from baseline to week 12 within group A and B.
   4. Comparison for the above mentioned parameters between group A and B. Treatment sessions will be for three months, daily oral cyclosporine and daily oral azathioprine and after completion, patients will be additionally followed for three more months.

      Oral cyclosporine 3mg/kg/day (200mg/day) will be started and given for one week, if patient shows improvement, the same dose will be continued for the total study period ( three months) ,after physical examination and various laboratory testing most importantly renal function tests, blood pressure monitoring, hemogram and if no symptomatic improvement then dose of cyclosporine will be increased slowly till 5 mg/kg /day.

      Oral azathioprine will be started at 1mg/kg/day ( 50mg/day) for one week , if patient demonstrates improvement, same dose is continued for the total study period ( 3months), after physical examination and various laboratory testing i.e LFTs, Hemogram, if no symptomatic improvement then dose of azathioprine will be increased to 2mg/kg/day (100mg/day).

      All the patients will be uniformly started on levocetrizine 10mg/day, which will continue daily for one month in all patients followed by stopping the drug and adding only if the patient is symptomatic.

      After three months both the drugs will be stopped and levocetrizine (10mg/day) will be continued for three months of follow up period.

      Clinical assessment of patients will be done before the starting of cyclosporine and azathioprine, and every fortnightly during three months of treatment and during three months of follow up period. Assessment will be done using UAS7and OSS as devised by Berroeta et al.

      URTICARIA ACTIVITY SCORE Table-2 SCORE WEALS PRURITUS

      0 None None

      1 Mild (<20 weals / 24 hours) Mild (present but not troublesome)

      2 Moderate (20-50 weals / 24 hours) Moderate (troublesome but does not interfere with sleep)

      3 Severe (>50 weals / 24 hours) Severe (sufficiently troublesome to interfere with normal daily activity and sleep)

      Scores of both parameters i.e. number of weals and severity of the pruritus per day are to be added to get UAS of that day and average UAS over 7 days is calculated which will range between 0 to 6. Patients will be instructed to write down number of weals and severity of itching in their daily urticaria diary. UAS7 will be calculated every fortnightly by calculating average of weal and itch score of the previous seven days after taking detailed history from patient.

      UAS7 SCORES71 HEALTH STATE

      0 Urticaria free

      1-6 Well controlled urticaria

      7-15 Mild urticaria

      16-27 Moderate urticaria

      26-42 Severe urticaria

      OUTCOME SCORING SCALE Another assessment scale i.e.Outcome scoring scale devised by Berroeta et al 22 for cyclosporine and azathioprine treatment of CU will also be used for clinical assessment of subjects.

      1- No change 2 - Minimal improvement (no change in frequency or extent, symptomatic improvement ±) 3- Moderate improvement (less frequent or extensive, symptomatic improvement +) 4- Marked improvement (occasional episodes and less extensive, symptomatic improvement ++) 5- Clearance

      In addition, ASST , APST and IgE levels will be done before starting cyclosporine and azathioprine and at the completion of the treatment after three months.

      FOLLOW UP After completion of oral cyclosporine and oral azathioprine for three months, patients will be followed up for a period of three more months, every fortnightly in urticaria clinic. At each visit, clinical assessment will be done using UAS7 and OSS. Urticaria being a type 1 hypersensitivity reaction, will relapse immediately as soon as the treatment is withheld. So, a follow up period of three months will be sufficient enough to study the effect of cyclosporine and azathioprine on long term remission of urticaria. Patients developing angioedema and having uncontrolled excessive exacerbation during treatment will be removed from study and will be treated accordingly.

      Patients who will fail to take the treatment for ≥ one week will be defined as defaulters and removed from the study. Those with no improvement even after one month of regular treatment will be labelled as non responders.

ELIGIBILITY:
Inclusion Criteria:

* Available definition for chronic refractory urticaria (CRU) is chronic spontaneous urticaria, with disease duration of at least 6 months or above, which is not controlled with four fold increased dosage of antihistamines (as per EAACI guidelines) figure1, given for at least three consecutive months and requiring repeated courses of oral corticosteroids.

Age ≥ 18 years.

Exclusion Criteria:

* Patients giving history of fainting, bronchospasm during previous attacks of urticaria that is suggestive of anaphylaxis.
* Urticaria< 6 weeks.
* Age <18 years.
* Physical and pressure urticaria.
* Urticarial vasculitits.
* Pregnant and lactating patients.
* Cataract, hepatic or renal diseases, severe infections, poorly controlled hypertension
* Concomitant intake of drugs like nephrotoxic drugs (gentamycin, vancomycin, amphotericin-B, indomethacin, diclofenac, H2 antihistamines like ranitidine, cimetidine, phenobarbitone, rifampicin, allupurinol, febuxostat).
* History suggestive of allergy to azathioprine , cyclosporine.
* Absolute contraindications69 of azathioprine are severe infections, severly impaired hepatic or bone marrow function, pancreatitis, live vaccines, pregnancy and lactation.
* Patients with chronic kidney disease, uncontrolled hypertension, renal insufficiency, uncontrolled infections, cutaneous T-cell lymphoma, including mycosis fungoides, should not be given Cyclosporine70.
* Patients who are planning pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in UAS7(urticaria activity score) ranging between( numerical value) 0-6 average of 7 days( primary end point) | 12 weeks
  Change in urticaria activity score (UAS7) ranging between 0-6 in average of 7 days i.e decrease more than 75% from baseline to week 12 (at end of treatment) within group A and B and comparison between corresponding groups.

SECONDARY OUTCOMES:
Change in OSS(outcome scoring scale) from baseline to 12 weeks ranging between( numerical value) 0-5 ( secondary end point) | 12 weeks
  a. Change in outcome scoring scale (OSS) ranging between 0-5 from baseline to week 12 within group A and B.
Change in ASST, APST( in milimeters),( numerical value) from baseline to week 12 within group A and B | 12 weeks
  Change in autologous serum and plasma skin tests measured in milimeters and considering its positivity and negativity within group A and B.
Change in S.IgE levels ( in UI/ml) from baseline to week 12 within group A and B | 12 weeks
  Change in serum IgE levels (in UI/ml) noted at baseline to week 12 within group A and B.
Change in both UAS7 and OSS ( secondary end point. | 24 weeks
  Change in UAS7 and OSS from baseline to week 24 (end of follow-up) within group A and B.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No